CLINICAL TRIAL: NCT04298307
Title: Prospective, Multicenter, Observational, Single-arm Registry of Coronary Lithotripsy for the Management of Calcified Lesions in Spain.
Brief Title: Registry of Coronary Lithotripsy in Spain.
Acronym: REPLICA
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC18-REPLICA
Record Dates: First submitted 2020-02-26; First posted 2020-03-06 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2022-07

CONDITIONS: Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Coronary Artery Disease
Keywords: Intracoronary lithotripsy; Calcified lesions; Percutaneous Coronary Intervention
MeSH Terms: conditions — Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with calcified coronary artery disease: Patients with calcified coronary artery disease require an ICL using the Shockwave catheter.
  Interventions: Other: Intracoronary lithotripsy (ICL)

INTERVENTIONS:
Other: Intracoronary lithotripsy (ICL) — ICL using the Shockwave catheter.

SUMMARY:
The REPLICA TRIAL tries to assess the intracoronary lithotripsy safety and efficacy profiles in real-world patients with calcified coronary artery disease.

DETAILED DESCRIPTION:
The REPLICA TRIAL tries to assess the intracoronary lithotripsy safety and efficacy profiles in real-world patients with calcified coronary artery disease requiring percutaneous revascularization with stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age.
* Patients with calcified coronary artery disease requiring percutaneous revascularization with stent implantation who, at the operator's discretion and according to the hospital routine clinical practice, require an ICL with the Shockwave catheter.
* The patients have been informed of the study characteristics and have given their written informed consent.

Exclusion Criteria:

* Refusal to participate in this study.
* Patients whose life expectancy is < 1 year.
* Patients with hemodynamic instability with Killip class III or IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be scheduled to undergo a intracoronary lithotripsy procedure using the Shockwave catheter (Shockwave Medical, Fremont, CA).
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Procedural success | Index Procedure
  Assessment of procedural success defined as angiographic results (TIMI grade 3 and residual stenosis < 20% without in-hospital complications ).

SECONDARY OUTCOMES:
MACE | Index Procedure
  Major Cardiovascular Adverse Events (MACE), defined as a composite of cardiac death, target vessel related nonfatal infarction or need for unplanned target vessel revascularization during hospital admission.
MACE | 12 months
  Major Cardiovascular Adverse Events (MACE), defined as a composite of cardiac death, target vessel related nonfatal infarction or need for unplanned target vessel revascularization.
Residual stenosis | Index Procedure
  Assessment of angiographic stenosis during stent implantation
Death (all cause) | 12 months
  Death (all cause)
Death (cardiovascular) | 12 months
  Death (cardiovascular)
Non-fatal Myocardial Infarction | 12 months
  Non-fatal Myocardial Infarction
Target Vessel Revascularization | 12 months
  Target Vessel Revascularization
Stent thrombosis of target lesion | 12 months
  Stent thrombosis of target lesion

CONTACTS AND LOCATIONS:
Locations (26):
- Spain (26):
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, Coruña
  - Hospital Universitario A Coruña, A Coruña, LA Coruña
  - Hospital Universitario Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario de Albacete, Albacete
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital de León, León
  - Hospital Universitario Lucus Agusti, Lugo
  - Hospital La Luz, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Central de La Defensa, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitari Joan Xxiii, Tarragona
  - Hospital Universitario Virgen de La Salud de Toledo, Toledo
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Universitario Miquel Servet, Zaragoza

REFERENCES:
- [Background] Brinton TJ, Ali ZA, Hill JM, Meredith IT, Maehara A, Illindala U, Lansky A, Gotberg M, Van Mieghem NM, Whitbourn R, Fajadet J, Di Mario C. Feasibility of Shockwave Coronary Intravascular Lithotripsy for the Treatment of Calcified Coronary Stenoses. Circulation. 2019 Feb 5;139(6):834-836. doi: 10.1161/CIRCULATIONAHA.118.036531. No abstract available. PMID 30715944
- [Background] Ali ZA, Nef H, Escaned J, Werner N, Banning AP, Hill JM, De Bruyne B, Montorfano M, Lefevre T, Stone GW, Crowley A, Matsumura M, Maehara A, Lansky AJ, Fajadet J, Di Mario C. Safety and Effectiveness of Coronary Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Stenoses: The Disrupt CAD II Study. Circ Cardiovasc Interv. 2019 Oct;12(10):e008434. doi: 10.1161/CIRCINTERVENTIONS.119.008434. Epub 2019 Sep 25. PMID 31553205
- [Background] Wong B, El-Jack S, Newcombe R, Glenie T, Armstrong G, Khan A. Shockwave Intravascular Lithotripsy for Calcified Coronary Lesions: First Real-World Experience. J Invasive Cardiol. 2019 Mar;31(3):46-48. doi: 10.25270/jic/19.00048. Epub 2019 Feb 15. PMID 30765621
- [Background] Vilalta V, Rodriguez-Leor O, Cid-Alvarez B, et al. Intracoronary Lithotripsy in a High-risk Real-world Population: First Experience in Severely Calcified, Complex Coronary Lesions. REC Interv Cardiol 2019; in press.
- [Background] Bourantas CV, Zhang YJ, Garg S, Iqbal J, Valgimigli M, Windecker S, Mohr FW, Silber S, Vries Td, Onuma Y, Garcia-Garcia HM, Morel MA, Serruys PW. Prognostic implications of coronary calcification in patients with obstructive coronary artery disease treated by percutaneous coronary intervention: a patient-level pooled analysis of 7 contemporary stent trials. Heart. 2014 Aug;100(15):1158-64. doi: 10.1136/heartjnl-2013-305180. Epub 2014 May 20. PMID 24846971
- [Derived] Rodriguez-Leor O, Cid-Alvarez AB, Lopez-Benito M, Gonzalo N, Vilalta V, Diarte de Miguel JA, Lopez LF, Jurado-Roman A, Diego A, Oteo JF, Cuellas C, Trillo R, Travieso A, Alfonso F, Carrillo X, Vegas-Valle JM, Cortes-Villar C, Pascual I, Munoz Camacho JF, Flores X, Vera-Vera S, Moreu J, Barreira de Sousa G, Marti D, Jimenez-Mazuecos J, Fuertes M, Ocaranza R, de la Torre Hernandez JM, Lozano F, Solana Martinez SG, Gomez-Lara J, Perez de Prado A; REPLICA-EPIC18 Investigators. A Prospective, Multicenter, Real-World Registry of Coronary Lithotripsy in Calcified Coronary Arteries: The REPLICA-EPIC18 Study. JACC Cardiovasc Interv. 2024 Mar 25;17(6):756-767. doi: 10.1016/j.jcin.2023.12.018. Epub 2024 Feb 21. PMID 38385926